CLINICAL TRIAL: NCT00005028
Title: Phase II Study of Weekly Paclitaxel and Bryostatin-1 in Hormone Refractory Prostate Cancer
Brief Title: Paclitaxel and Bryostatin 1 in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSGCC-9948; CDR0000067549 (Registry Identifier: PDQ (Physician Data Query)); NCI-50
Record Dates: First submitted 2000-04-06; First posted 2003-03-07 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bryostatin 1; Paclitaxel

ARMS (1):
- Arm I (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and bryostatin 1 IV over 1 hour on days 2, 9, and 16. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bryostatin 1; Drug: paclitaxel

INTERVENTIONS:
Drug: bryostatin 1
Drug: paclitaxel

SUMMARY:
Phase II trial to study the effectiveness of combining paclitaxel and bryostatin 1 in treating patients who have metastatic prostate cancer that has not responded to hormone therapy. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the onset, duration, and degree of response in patients with hormone-refractory, metastatic adenocarcinoma of the prostate treated with paclitaxel and bryostatin 1.

II. Determine the toxicity of this regimen in these patients. III. Determine the overall survival of patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and bryostatin 1 IV over 1 hour on days 2, 9, and 16. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly for 6 months and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic adenocarcinoma of the prostate that failed first- or second-line hormonal therapy (e.g., gonadal androgen suppression [orchiectomy or luteinizing hormone-releasing hormone] with or without antiandrogens)

  * Failure on hormonal therapy is defined by 1 of the following criteria:

    * Biochemical progression (after withdrawal of antiandrogens), documented by 3 rising PSA values, each value measured at least 2 weeks apart, with the last measurement being at least 25% of the nadir achieved while on hormonal therapy and with an increase in the absolute value by at least 5 ng/mL
    * Measurable disease progression, defined by an increase in the sum of the products of the perpendicular diameters of any measurable lesion(s) by at least 25%
* Bone only progression allowed only with concurrent biochemical progression
* Castrate levels of testosterone (no greater than 50 ng/dL)
* No clinical signs/symptoms suggesting CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 6 months

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN
* Calcium no greater than ULN

Cardiovascular

* No uncontrolled or severe cardiovascular disease
* No myocardial infarction within the past 6 months
* No congestive heart failure
* No angina pectoris
* No active thromboembolic events within the past 3 months (e.g., deep venous thrombosis or cerebrovascular accident)

Other

* No other serious medical or psychiatric illness
* No active infection
* No dementia or significantly altered mental status
* No prior or concurrent grade 1 or greater peripheral neuropathy
* No other prior or concurrent malignancy within the past 5 years except curatively treated nonmelanoma skin cancer
* HIV negative
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy (including paclitaxel)

Endocrine therapy

* At least 4 weeks since prior steroids or megestrol

Radiotherapy

* At least 4 weeks since prior radiotherapy to bone lesions

Other

* No other concurrent investigational therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2000-05 (Actual); Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arif Hussain, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (4):
- United States (4):
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Wellspan Health - York Cancer Center, York, Pennsylvania